CLINICAL TRIAL: NCT04541732
Title: Ultra-sound Guided Bilateral Quadratus Lumborum Block Versus Epidural Block for Postoperative Analgesia After Major Abdominal Surgeries.
Brief Title: Postoperative Analgesia of Quadratus Lumborum Block Versus Epidural Block After Major Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS ∕18.06.187
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Elective Major Abdominal Surgery
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Single blind study
Who Masked: Participant
Masking Description: Single blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural block (Experimental): Patients will receive thoracic epidural block following induction of general anaesthesia
  Interventions: Other: Thoracic epidural block; Drug: Induction of general anaesthesia with propofol; Drug: Muscle Relaxant; Drug: Maintenance of general anaesthesia
- Bilateral quadratus lumborum block (Active Comparator): Patients will receive Ultrasound-guided bilateral quadratus lumborum block following induction of general anaesthesia
  Interventions: Other: Ultrasound-guided bilateral quadratus lumborum block; Drug: Induction of general anaesthesia with propofol; Drug: Muscle Relaxant; Drug: Maintenance of general anaesthesia

INTERVENTIONS:
Other: Thoracic epidural block — Patients who will be subjected to epidural block will be placed in the lateral position then, after sterilization of the skin, 21 G spinal needle will be inserted at T9-T11 intervertebral spaces. The epidural space will be located using the loss of resistance to air technique and a mixture of bupivacaine 0.25% + 50 μ fentanyl targeting T6 level will be injected following induction of general anaesthesia.
  Arms: Thoracic epidural block
Other: Ultrasound-guided bilateral quadratus lumborum block — Patients who will be subjected to major abdominal surgeries will be placed in a supine position with a pillow under their side to obtain an appropriate view of quadratus lumborum muscle. After sterilization of the skin and ultrasound-guided identification of the quadratus lumborum muscle, 20 ml bupivacaine 0.25% + 25μ fentanyl will be injected on each side following induction of general anaesthesia
  Arms: Bilateral quadratus lumborum block
Drug: Induction of general anaesthesia with propofol — propofol: 1.5-2.5mg/Kg
Drug: Muscle Relaxant — Atracurium : 0.5mg/Kg.
Drug: Maintenance of general anaesthesia — Sevoflurane 0.7-1.5 MAC in 40% oxygen

SUMMARY:
Acute postoperative pain is an important issue after major abdominal surgeries for which different analgesic modalities have been tried.

Epidural analgesia is the recommended technique to relieve pain after major abdominal surgeries owing to the proved superior analgesia, reduction of opioid-related side effects as nausea, vomiting, pruritis and sedation, earlier recovery of bowel function and earlier ability for postoperative mobility. However, it is not without complications.

Quadratus lumborum block is an ultrasound-guided block that provides patients with both visceral and somatic blockade. It lessens the potential risks associated with neuraxial techniques, so it may represent a novel alternative approach for analgesia after major abdominal surgeries.

DETAILED DESCRIPTION:
The aim of this study is to detect the feasibility of ultra-sound guided bilateral quadratus lumborum block as a postoperative analgesic modality after major abdominal surgery in comparison to epidural block and its effects on total rescue analgesic requirements in the 1st postoperative 24hours, time to first analgesic request, pain VAS scores, intraoperative and postoperative hemodynamics and postoperative opioid-related side effects.

Under complete aseptic conditions, the patients will receive either thoracic epidural block or bilateral ultrasound-guided quadratus lumborum block after induction of general anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Patient's refusal
* Significant cardiac, disease.
* Significant hepatic disease.
* Significant renal disease (serum creatinine ˃ 1.5 mg/dl).
* Patients with drug abuse
* Allergy to study medications
* Mental disease
* Communication barrier.
* Coagulopathy.
* Local skin infection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Postoperative 24 hours cumulative rescue morphine consumption | For 24 hours after surgery

SECONDARY OUTCOMES:
The duration of postoperative analgesia | For 24 hours after surgery
  time from performing epidural or quadratus lumborum block till the time for the first rescue morphine request
Postoperative pain score at rest | For 24 hours after surgery
  Visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain)
Postoperative pain score on movement | For 24 hours after surgery
  Visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain)
Postoperative pain score on cough | For 24 hours after surgery
  Visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain)
Systolic blood pressure | For 28 hours after induction of anesthesia
Diastolic blood pressure | For 28 hours after induction of anesthesia
Mean blood pressure | For 28 hours after induction of anesthesia
Heart rate | For 28 hours after induction of anesthesia
Degree of postoperative nausea and vomiting | For 24 hours after surgery
  Nausea will be measured using a numerical rating system (none= 0; mild= 1; moderate= 2; severe= 3). The number of vomiting episodes and the number of antiemetics received will be recorded
Pruritis | For 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Ghanem, MD, Study Director — Associate Professor; Mona A Hasheesh, MD, Study Chair — Professor
Locations (1):
- Mohammed A Ghanem, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided